CLINICAL TRIAL: NCT01053533
Title: A Pragmatic Randomized Controlled Trial of Chinese Herbal Medicine for Severe Pandemic H1N1 Influenza
Acronym: 200907001-2A
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Collaborators: Beijing University of Chinese Medicine (Other); State Administration of Traditional Chinese Medicine of the People's Republic of China (Other Government); China Academy of Chinese Medical Sciences (Other)
Responsible Party: Beijing Di Tan Hospital, Beijing Di Tan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20100118
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-01

CONDITIONS: Influenza A Virus, H1N1 Subtype
Keywords: Chinese herbal medicines; pandemic H1N1 influenza; effectiveness; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese herbal medicines plus western therapy (Experimental)
  Interventions: Drug: Chinese herbal medicines plus western therapy
- western therapy (Active Comparator): including supportive therapy and antivirus therapy when necessary
  Interventions: Drug: western therapy

INTERVENTIONS:
Drug: Chinese herbal medicines plus western therapy — injections of Chinese herbal medicines and Chinese herbal medicines decoction& supportive therapy and antivirus therapy when necessary
  Arms: Chinese herbal medicines plus western therapy
Drug: western therapy — supportive therapy and antivirus therapy when necessary
  Arms: western therapy

SUMMARY:
The aim of this study is to evaluate the effectiveness and safety of Chinese herbal medicines for severe pandemic H1N1 influenza.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of severe pandemic H1N1 influenza patients and pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza
* Rapid Diagnostic Tests:positive
* Age≥6 years
* Influenza symptoms occurred less than 48 hours and body temperature≥37.5℃ for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza

Exclusion Criteria:

* Suffering from mental illness
* Attending other clinical studies on influenza
* Critical pandemic H1N1 influenza patients

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
incidence of complication | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients.
mortality of pandemic H1N1 influenza and all-cause mortality(only for severe pandemic H1N1 influenza patients) | 28 days
proportion of deteriorating into severe H1N1 influenza (only for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza) | 10 days

SECONDARY OUTCOMES:
time to allaying a fever | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
time to symptom relief | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
time and proportion of H1N1 virus turning to negative | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
direct medical cost | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
safety outcome(adverse effects) | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
days in hospital | 10 days for pandemic H1N1 influenza patients with risk factors for severe H1N1 influenza;28 days for severe pandemic H1N1 influenza patients
dose and usage of hormones(only for severe pandemic H1N1 influenza patients) | 28 days
Inflammation of lung tissue(only for severe pandemic H1N1 influenza patients) | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Mao Yu, Beijing, Beijing Municipality, China